CLINICAL TRIAL: NCT00830323
Title: Efficacy and Safety of Combination Therapies With Oseltamivir & Zanamivir or Oseltamivir & Amantadine Versus Oseltamivir Monotherapy in the Treatment of Seasonal Influenza A Infection
Acronym: Combina
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Pr Bruno LINA, Laboratoire de Virologie/Centre de Biologie et de Pathologie EST
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-517
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2009-10

CONDITIONS: Influenza A Infection
MeSH Terms: interventions — Oseltamivir; Zanamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: oseltamivir + zanamivir
- Arm 2 (Experimental)
  Interventions: Drug: oseltamivir+ amantadine
- Arm 3 (Active Comparator)
  Interventions: Drug: oseltamivir

INTERVENTIONS:
Drug: oseltamivir + zanamivir — oseltamivir (75mg bd for 5 days, oral) zanamivir (5mg bd for 5 days, inhaled by mouth)
  Arms: 1
Drug: oseltamivir+ amantadine — oseltamivir (75mg bd for 5 days, oral) + amantadine (100mg bd for 5 days, oral)
  Arms: Arm 2
Drug: oseltamivir — oseltamivir (75mg bd for 5 days, oral)
  Arms: Arm 3

SUMMARY:
Neuraminidase inhibitors (NAI) are effective anti-influenza antiviral treatment. During their use in experimentally infected patients, it has been shown that the viral load detected in the nasal fluid is decreasing significantly faster than in non treated patients. During clinical practice, the emergence of NAI-resistant strains has been observed. These strains remain rare, but their emergence seemed to be related to the mis-use of the NAI products (insufficient duration or dosage). This observation as well as the detection of NAI-resistant viruses in the community raises concerns about putative emergence of resistant clones in the specific context of a pandemic, when the use of NAI will be very large in the aim of reducing transmission, and subsequently the impact of the emerging virus.

In this context, it is important to determine the putative interest of alternative strategies.

Although zanamivir and oseltamivir are both issued from the same class , this combination may lead to a more rapid viral clearance in the infected cases, and to a reduction in the emergence of resistant sub-clones, and alternatively, might lead to a competitive inhibition. The evaluation of these combinations needs to be conducted in vivo.

Among available anti influenza antivirals, M2 blockers have been previously used. Although their efficacy against A H5N1 remains to be ascertained, their use in combination with NAI should also be evaluated in the context of a preparation for a possible pandemic and determination of the stockpile.

Therefore, the evaluation of combination therapies in the treatment of a virologically suspected influenza will be investigated in primary care during the winter season 2008-2009.

DETAILED DESCRIPTION:
Study Schedule:

* Patient's follow up: 7 days with 10 visits V1, V2, V3, V4, V5 every 12 hours V6, V7, V8, V9, V10 every 24 hours
* V1: conducted by the GP rapid test diagnostic for influenza A, urine pregnancy test for women, inclusion /randomisation, nasal sample, initiation of treatment.
* V2 to V9: conducted by a nurse at the patient's home; nasal sample, symptoms scoring, safety assessment (side effects)
* V 10: conducted by GP; medical evaluation (follow up evaluation)

ELIGIBILITY:
Inclusion Criteria:

* Influenza season declared
* Subjects aged>18 years and < 65 years presenting within 36h documented of onset influenza illness
* Who have fever >38°C
* Who present at least one of the following respiratory symptoms (cough, sore throat, nasal symptoms), and one of the following constitutional symptoms (headache, myalgia, sweats and or chills or fatigue)
* Positive rapid diagnostic test for influenza A
* Who have giving written informed consent prior to enrollment
* Patient examined before the inclusion
* Primary care follow up

Exclusion Criteria:

* Influenza Vaccination in the 12 months prior the beginning of the study
* Asthma, Chronic bronchitis
* Woman with a positive urine pregnancy test
* Active breast feeding
* Woman without contraception
* Clearance of creatinine< 30 ml/min Chronic renal disease
* History of depression, psychiatric disorders, epilepsy
* Patients receiving cortocosteroids, immunosuppressants or antipsychotic antiemetic drugs
* Known oseltamivir or zanamivir hypersensibility
* Non member of the social security or CMU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
describe the antiviral efficacy in the 3 arms in the treatment of seasonal influenza infection as assessed by negative viral detection in nose swabs at the fifth swab [H48±3] | 48 hours
Describe the antiviral efficacy in 3 arms in the treatment of seasonal influenza infection as assessed by negativity of RT-PCR for viral RNA in nose and throat swabs at the 5th swab [H48±3] and at the 7th swab [H84±3]. | 84 hours

SECONDARY OUTCOMES:
Describe the antiviral efficacy in combination therapy arms (1,2) and in monotherapy arm (3) in the treatment of seasonal influenza infection as assessed by time to sustained negativity of RT-PCR for viral RNA or viral culture in any sample. | 168 hours
Assess viral replication dynamics (duration and level of viral replication) in the respiratory tract in the combination and standard-dose cohorts. | 168 hours
Assess the frequency, genetic basis, and duration of antiviral resistance to each arm during and after therapy | 168 hours
Describe the time to alleviation of illness in the 3 arms defined as the time from the beginning of the study treatment to the time that 7 typical key symptoms of natural influenza had reduced to absent or mi | 168 hours
Describe the tolerability of combination and in standard-dose arms as assessed by clinical adverse events that are possibly or probably related to each single agent (Incidence and duration) | 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: BRUNO LINA, MD,PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices civils de Lyon, Lyon, France